CLINICAL TRIAL: NCT01962909
Title: A Phase 0, Open Label Study to Evaluate the Biodistribution and Pharmacokinetics of a Single Intravenous Bolus Dose of PTP-01 in Subjects With Resectable Pancreatic Ductal Adenocarcinoma
Brief Title: Phase 0 Biodistribution of Novel Imaging for Resectable Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: From preliminary imaging data, the study was stopped due to futility.
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16678
Record Dates: First submitted 2013-06-19; First posted 2013-10-14 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PTP-01 (Experimental): single IV bolus dose 24 hours prior to surgery
  Interventions: Drug: PTP-01

INTERVENTIONS:
Drug: PTP-01 — Dose level 1 is 10mCi (50ug of peptide)

SUMMARY:
The purpose of this clinical trial is to study an experimental drug called PTP-01 that is being used as an imaging agent to diagnosis pancreatic cancer. Currently, pancreatic cancer is diagnosed using CT or MRI scans which miss small pancreatic cancers, particularly early stage disease. Researchers at the University of Virginia have identified a biomarker for pancreatic cancer called plectin, which is very specific for pancreatic cancer and not other, non-cancerous conditions involving the pancreas. These researchers have also developed PTP-01, an experimental drug that may be used with SPECT imaging to detect pancreatic cancer cells in humans.

ELIGIBILITY:
Inclusion Criteria:

* subject is undergoing resection of pancreas for pancreatic ductal adenocarcinoma (PDAC)
* subject must have adequate renal function
* ECOG performance status of 0-2
* women of child-bearing age and men must agree to use contraception prior to and during the study

Exclusion Criteria:

* subjects receiving any other investigational agents
* significant history of uncontrolled cardiac disease or central nervous system (CNS) disease
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Ability of PTP-01 to detect pancreatic ductal adenocarcinoma | up to 72 hours post dose
  requires a signal to background ratio of greater than or equal to 2:1 following a single intravenous bolus of PTP-01

SECONDARY OUTCOMES:
Biodistribution and Binding Characteristics of PTP-01 | up to 7 days post dose
  Assessments will be made from imaging (whole body planar and SPECT/CT) and blood draws following PTP-01 dose. Tissue samples will also be retained for pathology.
Clearance of PTP-01 | up to 7 days post dose
  Blood and urine samples will be collected to measure the level of radioactivity at specified intervals following PTP-01 dose.
Safety and Tolerability of PTP-01 | up to 30 days post dose
  Clincial labs, ECGs, vital signs and physical exams will be performed up to 7 days post dose. Adverse events will be collected up to 30 days post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Reid Adams, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States